CLINICAL TRIAL: NCT00778713
Title: A Bioequivalence Study of Test and Reference Fosinopril Sodium/ Hydrochlorothiazide 20/ 12.5 mg Tablets Under Non-Fasting Conditions
Brief Title: Bioequivalence Study of Fosinopril Sodium / Hydrochlorothiazide 20/ 12.5 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B035502
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Fosinopril; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets of Ranbaxy laboratories Limited
  Interventions: Drug: Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets
- 2 (Active Comparator): Monopril ® - HCT 20-12.5 mg tablets by Bristol Meyers Squibb following a single oral dose (1 x 20/12.5 mg tablet)
  Interventions: Drug: Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets

INTERVENTIONS:
Drug: Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets

SUMMARY:
The objective of this study is to compare the relative bioavailability of Fosinopril sodium and hydrochlorothiazide 20-12.5 mg tablets of Ranbaxy laboratories Limited with that of Monopril ® - HCT 20-12.5 mg tablets by Bristol Meyers Squibb following a single oral dose (1 x 20/12.5 mg tablet) in healthy adult subjects under non-fasting conditions.

DETAILED DESCRIPTION:
This study was a single dose, randomized, two-period, two-sequence, crossover design study. It was used to evaluate the relative bioavailability of the Fosinopril sodium and hydrochlorothiazide tablet products when dose (1 x 20/ 12.5 mg) under non-fasting conditions. There was a washout of at least a week between the two study periods.

A total of thirty six (36) healthy adult volunteers were recruited in the study of which only thirty three (33) subjects i.e. 18 males and 15 females completed the clinical portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should be at least 18 years old
2. Female subjects with negative serum pregnancy test
3. Subject with no clinically significant abnormal lab values at the pre-entry evaluation
4. Subjects with negative or non-reactive urine drug of abuse, hepatitis B, hepatitis C and HIV screening
5. Subject has acceptable ECG
6. Subject has no evidence of underlying disease at the pre-entry physical examination
7. Subject has agreed to undergo at least a 14 day washout period for prescription drugs prior to the first dosing of the study and throughout the periods of blood sample collection
8. Subject has agreed to undergo at least a 7 day washout period for OTC products, herbal medications, etc. prior to the first dosing of the study medication and throughout the periods of blood sample collections
9. Subject agrees to abstain from consuming alcohol for at least 48 hours prior to each dosing and throughout the periods when blood samples are being obtained
10. Subject agrees to abstain from consuming grapefruit, grapefruit juice, or other foods containing grapefruit for at least 48 hours prior to each dosing and throughout the periods when blood samples are being obtained
11. Subject has given a written consent to participate

Exclusion Criteria:

1. Subject has a history of chronic alcohol consumption (during past 2 years) or drug addiction
2. Subject has a history of serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma
3. Subject has a history of allergic responses to the class of drug being tests
4. Subject has donated any blood and/ or plasma within the last thirty (30) days prior to the first dosing of the study
5. Subject has taken any investigational drug within thirty (30) days prior to the first dosing of the study
6. Female subjects who are pregnant, breast feeding, or likely to be come pregnant during the study. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (eg condom, IUD) of contraception during the course of the study (first dosing until the last blood collection)
7. Female subjects who have used implanted or injected hormonal contraceptives (except Lunelle ® Monthly Injection) anytime during the 6 months prior to study dosing, Lunelle ® Monthly Injection anytime during the 45 days prior to the study dosing, or used oral hormonal contraceptives within 14 days before dosing.
8. Subject with the inability to read and/ or sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-03; Primary Completion 2003-03 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Medical Research Inc, Saint Charles, Missouri, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html